CLINICAL TRIAL: NCT00029510
Title: Magnesium and Asthma - Clinical Trials
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000652-02 (NIH)
Record Dates: First submitted 2002-01-14; First posted 2002-01-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Magnesium

INTERVENTIONS:
Drug: Magnesium

SUMMARY:
Asthma currently affects an estimated 15 million Americans. A number of studies have found an association between low dietary magnesium (Mg) intake and increased asthma incidence and severity of symptoms. However, clinical intervention trials are necessary to directly assess whether there is a true protective or preventative causal relationship between low Mg and asthma. In our study, we will assess the effects of 6 1/2 months of oral Mg supplements or placebo on clinical markers of asthma control, indirect biomarkers of inflammation, bronchial hyperresponsiveness, and indices of oxidative defense and damage in subjects with mild to moderate persistent asthma.

DETAILED DESCRIPTION:
Over the past twenty years a number of studies of acute bronchial asthma have shown that i.v. or nebulized MgS04 may improve symptoms over a course of hours. With respect to dietary supplementation, short term (3 wk) oral Mg has been associated with a significant decrease in symptoms but no significant effect on measurements like FEV1 or bronchial hyperreactivity by methacholine challenge. Although a large number of studies have attempted to address this issue, we believe that major gaps still exist. One of the gaps is in the comparison of large numbers of asthmatics and non-asthmatics, with regard to dietary intake, and a variety of measures of Mg status. We will evaluate baseline Mg intake (diet, tap and bottled drinking water, vitamin-mineral supplements, laxatives, and antacids), and multiple measures of Mg status, such as total and free serum Mg, total erythrocyte Mg, and Mg retention after an IV Mg load in subjects with and without asthma. Furthermore there are no large-scale studies evaluating the effects of Mg supplementation on asthma control and clinical markers, and markers of inflammation. We propose to assess the effects of 6 1/2 months of oral Mg on clinical markers of asthma control (asthma symptom diary, monthly spirometry, asthma quality of life questionnaire (QOL)), indirect biomarkers of inflammation (exhaled nitric oxide and serum eosinophil cationic protein) and bronchial hyperresponsiveness (methacholine challenge)in subjects with mild to moderate persistent asthma. Dietary Mg will be assessed using the 24 hr recall. Our hypotheses are that 1.) subjects with mild to moderate persistent asthma, as defined by National Institutes of Health National Asthma Education and Prevention Program (NIH NAEPP) clinical guidelines will have poorer Mg status than nonasthmatics, and 2.) that marginal Mg intake and status may modulate the severity of asthma. Thus, subjects with asthma who have marginal intake/status and thus relatively lower total and free plasma Mg, lower erythrocyte total Mg, and higher Mg retention will show improvement in the aforementioned clinical and indirect biomarkers. In contrast, Mg supplements will have little effect in subjects with highest intakes and Mg status. We do not anticipate that Mg supplementation will replace conventional treatment, but may complement and decrease the need for conventional medication.

ELIGIBILITY:
* Mild to moderate persistent asthma (NAEPP 1997 revised guidelines)
* Current use of inhaled beta-2- agonists or steroid inhaler therapy only (No use of prednisone in past 3 months)
* No use of products (i.e. antacids, laxatives, supplements) containing more than 50 mg Mg daily in the last 3 months
* No current use of theophylline, leukotriene antagonists, or other systemic immunomodulating compounds
* Nonsmoker
* No concurrent pulmonary disease (pulmonary hypertension, cystic fibrosis, sarcoidosis, bronchiectasis, hypersensitivity pneumonitis, restrictive lung disease, abnormal DLCOva)
* No concurrent medical diagnoses (alcoholism, coronary artery disease, diabetes, HIV infection, chronic hepatitis, uncontrolled hypertension, chronic renal failure or a psychiatric disorder that is judged to make full participation difficult)
* Not pregnant or lactating.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240
Dates: Start 2002-05; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Stern, Sc.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California at Davis School of Medicine, Ticon 1, Suite 100B, 2000 Stockton Blvd, Sacramento, California, United States

REFERENCES:
- [Derived] Kazaks AG, Uriu-Adams JY, Albertson TE, Shenoy SF, Stern JS. Effect of oral magnesium supplementation on measures of airway resistance and subjective assessment of asthma control and quality of life in men and women with mild to moderate asthma: a randomized placebo controlled trial. J Asthma. 2010 Feb;47(1):83-92. doi: 10.3109/02770900903331127. PMID 20100026